CLINICAL TRIAL: NCT03996291
Title: Long-term Extension Safety and Efficacy Study of SAR442168 in Participants With Relapsing Multiple Sclerosis
Brief Title: Long Term Safety and Efficacy Study of Tolebrutinib (SAR442168) in Participants With Relapsing Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTS16004; U1111-1223-4256 (Registry Identifier: ICTRP); 2018-004731-76 (EudraCT Number)
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Results first posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Relapsing Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SAR442168 (Experimental): SAR442168 : Experimental - Part A: Double-blind period of continued treatment with the respective SAR442168 dose was administered in the DRI15928 study until selection of Phase 3 dose.
  Part B: Open-label period of a single-group treatment with SAR442168 selected Phase 3 dose of 60 mg. All participants were switched to this 60 mg dose.
  Interventions: Drug: Tolebrutinib

INTERVENTIONS:
Drug: Tolebrutinib — Pharmaceutical form: Film coated tablet Route of administration: Oral
  Other Names: SAR442168

SUMMARY:
Primary Objective:

To determine the long-term safety and tolerability of SAR442168 in RMS participants

Secondary Objective:

To evaluate efficacy of SAR442168 on disease activity, assessed by clinical and imaging methods

DETAILED DESCRIPTION:
Approximately 62 months including the 8 weeks post-treatment visit

ELIGIBILITY:
Inclusion criteria:

* Participants had to have completed treatment in the DRI15928 study
* Female participants had to continue to use an acceptable effective contraception method of birth control from inclusion and until the last dose of study drug, except if she had undergone sterilization at least 3 months earlier or was postmenopausal. Menopause was defined as being amenorrheic for ≥12 months with plasma follicle stimulating hormone (FSH) level >30 UI/L.
* The participant had to have given written informed consent prior to undertaking any study related procedure.

Exclusion criteria:

* The participant had a confirmed concomitant laboratory or ECG abnormality or medical condition deemed by the investigator incompatible with continuation of SAR442168 treatment.
* The participant had received any live (attenuated) vaccine (including but not limited to varicella zoster, oral polio, and nasal influenza) between the last DRI15928 visit and the first treatment visit in the LTS16004 study.
* The participant had received a non-study MS disease modifying treatment between the last IMP treatment in Study DRI15928 and inclusion in Study LTS16004, which by judgement of the Investigator may add unjustified risk to switching back and continuing treatment with SAR442168. Washout periods after treatment with non-study DMTs had to be respected except for interferons or glatiramer acetate treatment.
* The participant was receiving strong inducers or inhibitors of CYP3A or CYP2C8 hepatic enzymes.
* The participant was receiving anticoagulant/antiplatelet therapies, including:

  * Acetylsalicylic acid (aspirin)
  * Antiplatelet drugs (eg, clopidogrel)
  * Warfarin (vitamin K antagonist)
  * Heparin, including low molecular weight heparin (antithrombin agents)
  * Dabigatran (direct thrombin inhibitor)
  * Apixaban, edoxaban, rivaroxaban (direct factor Xa inhibitors)

Note: All above drugs needed to be stopped at least 5 half-lives before study drug administration except for aspirin, which needed to be stopped at least 8 days beforehand.

* Prior/concurrent clinical study experience. The participant was taking part in another interventional clinical trial of another drug substance.
* Uncooperative behavior or any condition that could make the participant potentially non-adherent with the study procedures
* The participant was pregnant or was a breastfeeding woman.

The above information was not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (37):
- United States (8):
  - North Central Neurology Associates, PC Site Number : 8400005, Cullman, Alabama
  - Neurology Associates, PA Site Number : 8400002, Maitland, Florida
  - University of South Florida Site Number : 8400009, Tampa, Florida
  - Velocity Clinical Research Site Number : 8400007, Savannah, Georgia
  - Consultants In Neurology Site Number : 8400001, Northbrook, Illinois
  - UC Health, LLC Site Number : 8400008, Dayton, Ohio
  - MDH Research LLC Site Number : 8400006, Westerville, Ohio
  - Neurology PC Site Number : 8400003, Knoxville, Tennessee
- Canada (2):
  - Investigational Site Number : 1240003, Vancouver, British Columbia
  - Investigational Site Number : 1240001, Greenfield Park, Quebec
- Czechia (7):
  - Investigational Site Number : 2030007, Brno
  - Investigational Site Number : 2030004, Hradec Králové
  - Investigational Site Number : 2030003, Jihlava
  - Investigational Site Number : 2030005, Ostrava - Poruba
  - Investigational Site Number : 2030006, Pardubice
  - Investigational Site Number : 2030001, Prague
  - Investigational Site Number : 2030002, Praha 5 - Motol
- Investigational Site Number : 2330001, Tallinn, Estonia
- Investigational Site Number : 2500004, Nancy, France
- Investigational Site Number : 5280001, Amsterdam, Netherlands
- Russia (5):
  - Investigational Site Number : 6430006, Kazan'
  - Investigational Site Number : 6430003, Moscow
  - Investigational Site Number : 6430005, Saint Petersburg
  - Investigational Site Number : 6430001, Saint Petersburg
  - Investigational Site Number : 6430007, Tyumen
- Spain (5):
  - Investigational Site Number : 7240003, Seville, Andalusia
  - Investigational Site Number : 7240002, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240005, Salt, Girona [Gerona]
  - Investigational Site Number : 7240001, Madrid
  - Investigational Site Number : 7240004, Murcia
- Ukraine (7):
  - Investigational Site Number : 8040002, Chernivtsi
  - Investigational Site Number : 8040005, Dnipro
  - Investigational Site Number : 8040001, Lviv
  - Investigational Site Number : 8040006, Lviv
  - Investigational Site Number : 8040009, Odesa
  - Investigational Site Number : 8040003, Vinnytsia
  - Investigational Site Number : 8040007, Zhytomyr

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LTS16004 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25300&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This long-term study was conducted at 37 centers in 9 countries. Of the 129 participants who completed the parent study DRI15928 (NCT03889639), 126 were screened in this study from 23-Sep-2019 to 10-Mar-2020 of which 1 failed screening due to not meeting eligibility criteria.
Pre-assignment Details: A total of 125 participants were treated in this study which consisted of 2 parts: Part A (double-blind) and Part B (open-label). Part A was a short transition period until the dose of tolebrutinib to be used in Phase 3 was determined. In Part B, all participants formed a single dose group (the selected Phase 3 dose).
Groups:
- Part A: Tolebrutinib 5 mg: Participants who received tolebrutinib 5 milligrams (mg) orally once daily in the parent study continued to receive the same dose until the dose of tolebrutinib to be used in Phase 3 was determined.
- Part A: Tolebrutinib 15 mg: Participants who received tolebrutinib 15 mg orally once daily in the parent study continued to receive the same dose until the dose of tolebrutinib to be used in Phase 3 was determined.
- Part A: Tolebrutinib 30 mg: Participants who received tolebrutinib 30 mg orally once daily in the parent study continued to receive the same dose until the dose of tolebrutinib to be used in Phase 3 was determined.
- Part A: Tolebrutinib 60 mg: Participants who received tolebrutinib 60 mg orally once daily in the parent study continued to receive the same dose until the dose of tolebrutinib to be used in Phase 3 was determined.
- Part B: Tolebrutinib 5/60 mg: Participants from Part A: tolebrutinib 5 mg arm who provided consent switched to Part B to receive the selected Phase 3 dose of tolebrutinib 60 mg orally once daily until Month 60.
- Part B: Tolebrutinib 15/60 mg: Participants from Part A: tolebrutinib 15 mg arm who provided consent switched to Part B to receive the selected Phase 3 dose of tolebrutinib 60 mg orally once daily until Month 60.
- Part B: Tolebrutinib 30/60 mg: Participants from Part A: tolebrutinib 30 mg arm who provided consent switched to Part B to receive the selected Phase 3 dose of tolebrutinib 60 mg orally once daily until Month 60.
- Part B: Tolebrutinib 60/60 mg: Participants from Part A: tolebrutinib 60 mg arm who provided consent switched to Part B and continued to receive the selected Phase 3 dose of tolebrutinib 60 mg orally once daily until Month 60.
Period: Part A (Double-blind Period):39 Weeks
Arm/Group | Part A: Tolebrutinib 5 mg | Part A: Tolebrutinib 15 mg | Part A: Tolebrutinib 30 mg | Part A: Tolebrutinib 60 mg | Part B: Tolebrutinib 5/60 mg | Part B: Tolebrutinib 15/60 mg | Part B: Tolebrutinib 30/60 mg | Part B: Tolebrutinib 60/60 mg
Started (Treated) | 31 | 31 | 32 | 31 | 0 | 0 | 0 | 0
Completed | 30 | 31 | 32 | 31 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B (Open-label Period):222 Weeks
Arm/Group | Part A: Tolebrutinib 5 mg | Part A: Tolebrutinib 15 mg | Part A: Tolebrutinib 30 mg | Part A: Tolebrutinib 60 mg | Part B: Tolebrutinib 5/60 mg | Part B: Tolebrutinib 15/60 mg | Part B: Tolebrutinib 30/60 mg | Part B: Tolebrutinib 60/60 mg
Started (All participants who completed Part A and provided consent switched to Part B.) | 0 | 0 | 0 | 0 | 30 | 31 | 32 | 31
Completed | 0 | 0 | 0 | 0 | 20 | 23 | 20 | 26
Not Completed | 0 | 0 | 0 | 0 | 10 | 8 | 12 | 5
Not completed — Poor compliance to protocol | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 8 | 7 | 10 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all participants enrolled in this study and exposed to study drug, regardless of the amount of exposure.
Groups:
- Part A: Tolebrutinib 5 mg: Participants who received tolebrutinib 5 mg orally once daily in the parent study continued to receive the same dose until the dose of tolebrutinib to be used in Phase 3 was determined.
- Total: Total of all reporting groups
Arm/Group | Part A: Tolebrutinib 5 mg | Part A: Tolebrutinib 15 mg | Part A: Tolebrutinib 30 mg | Part A: Tolebrutinib 60 mg | Total
Number analyzed (Participants) | 31 | 31 | 32 | 31 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (9.9) | 36.4 (9.4) | 40.0 (9.9) | 37.8 (9.0) | 37.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 20 | 23 | 86
  Male | 8 | 11 | 12 | 8 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 2 | 6
  White | 30 | 29 | 28 | 28 | 115
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study drug, whether or not considered related to the study drug. An SAE was any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, was a congenital anomaly/birth defect or was an important medical event. TEAEs were defined as AEs that developed, worsened or became serious during the respective on-treatment periods.
Time Frame: From first dose of study drug (Day 1) up to maximum exposure, 39 weeks in Part A and 222 weeks in Part B
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Tolebrutinib 5 mg | Part A: Tolebrutinib 15 mg | Part A: Tolebrutinib 30 mg | Part A: Tolebrutinib 60 mg | Part B: Tolebrutinib 5/60 mg | Part B: Tolebrutinib 15/60 mg | Part B: Tolebrutinib 30/60 mg | Part B: Tolebrutinib 60/60 mg
Number analyzed (Participants) | 31 | 31 | 32 | 31 | 30 | 31 | 32 | 31
Participants
  TEAEs | 17 | 17 | 24 | 20 | 26 | 29 | 27 | 27
  TESAEs | 0 | 2 | 1 | 2 | 5 | 3 | 3 | 3

2. Secondary Outcome: Mean Number of New Gadolinium (Gd)-Enhancing T1-hyperintense Lesions at Week 240 Relative to Week 192
Description: Magnetic resonance imaging (MRI) of the brain was performed to identify number of new Gd-enhancing T1-hyperintense lesions. Central review was used to identify new Gd-enhancing T1-hyperintense lesions not present at the previous MRI. mITT=modified intent-to-treat; SAP= statistical analysis plan. Only those participants with data collected at specified timepoints are reported.
Time Frame: Weeks 192 and 240
Population: The mITT population included all participants enrolled in this study who had at least 1 day of study drug exposure during study. As pre-specified in protocol and SAP, the main objective of this study was to determine the long-term efficacy of selected Phase 3 dose (60 mg). Part A was a short transition period while picking phase 3 dose; no efficacy analysis was planned for this period alone. Hence, complete efficacy data is presented by LTS16004 dose groups of 5/60, 15/60, 30/60 and 60/60 mg.
Measure: Mean (Standard Deviation); unit: number of new Gd-enhancing T1 lesions
Groups:
- Tolebrutinib 5/60 mg: All participants who received tolebrutinib 5 mg in Part A and tolebrutinib 60 mg in Part B were included in this arm.
- Tolebrutinib 15/60 mg: All participants who received tolebrutinib 15 mg in Part A and tolebrutinib 60 mg in Part B were included in this arm.
- Tolebrutinib 30/60 mg: All participants who received tolebrutinib 30 mg in Part A and tolebrutinib 60 mg in Part B were included in this arm.
- Tolebrutinib 60/60 mg: All participants who received tolebrutinib 60 mg in Part A and tolebrutinib 60 mg in Part B were included in this arm.
Arm/Group | Tolebrutinib 5/60 mg | Tolebrutinib 15/60 mg | Tolebrutinib 30/60 mg | Tolebrutinib 60/60 mg
Number analyzed (Participants) | 21 | 22 | 19 | 24
number of new Gd-enhancing T1 lesions | 0.24 (0.54) | 0.36 (0.66) | 0.32 (0.75) | 0.13 (0.45)

3. Secondary Outcome: Mean Number of New or Enlarging T2 Lesions at Week 240 Relative to Week 192
Description: MRI of the brain was performed to identify number of new or enlarging T2 lesions. Central review was used to identify new or enlarging T2 lesions not present at the previous MRI; the values were standardized to per month values by dividing by the number of months (4-week intervals) from the previous MRI to the current MRI.
Time Frame: Weeks 192 and 240
Population: Analysis was performed on the mITT population. As pre-specified in protocol and SAP,main objective of this study was to determine long-term efficacy of selected Phase 3 dose (60 mg).Part A was a short transition period while picking phase 3 dose;no efficacy analysis was planned for this period alone. Hence, complete efficacy data is presented by LTS16004 dose groups of 5/60, 15/60, 30/60, and 60/60 mg. Only those participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: new or enlarging T2 lesions/month
Arm/Group | Tolebrutinib 5/60 mg | Tolebrutinib 15/60 mg | Tolebrutinib 30/60 mg | Tolebrutinib 60/60 mg
Number analyzed (Participants) | 21 | 23 | 21 | 26
new or enlarging T2 lesions/month | 0.32 (0.54) | 0.37 (0.53) | 0.15 (0.30) | 0.24 (0.41)

4. Secondary Outcome: Total Mean Number of Gd-enhancing T1-hyperintense Lesions at Week 240 Relative to Week 192
Description: MRI of the brain was performed to identify number of Gd-enhancing T1-hyperintense lesions. Central review was used to identify Gd-enhancing T1-hyperintense lesions not present at the previous MRI.
Time Frame: Weeks 192 and 240
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: number of Gd-enhancing T1 lesions
Arm/Group | Tolebrutinib 5/60 mg | Tolebrutinib 15/60 mg | Tolebrutinib 30/60 mg | Tolebrutinib 60/60 mg
Number analyzed (Participants) | 21 | 22 | 19 | 24
number of Gd-enhancing T1 lesions | 0.24 (0.54) | 0.36 (0.66) | 0.37 (0.76) | 0.13 (0.45)

5. Secondary Outcome: Annualized Relapse Rate (ARR)
Description: Multiple sclerosis (MS) relapse was defined as acute, new neurological symptoms or worsening of previous neurological symptoms with an objective change on neurological examination. Symptoms were attributable to MS, lasted for >=24 hours with or without recovery, present at normal body temperature and preceded by >=30 days of clinical stability. ARR was the total number of relapses for participants by dose group divided by the sum of the standardized study duration for participants in the dose group.
Time Frame: From Baseline (enrollment in LTS16004, Day 1) to Week 240
Population: Analysis was performed on the mITT population. As pre-specified in protocol and SAP,main objective of this study was to determine long-term efficacy of selected Phase 3 dose (60 mg).Part A was a short transition period while picking phase 3 dose;no efficacy analysis was planned for this period alone. Hence, complete efficacy data is presented by LTS16004 dose groups of 5/60, 15/60, 30/60, and 60/60 mg.
Measure: Number (95% Confidence Interval); unit: relapses per participant year
Arm/Group | Tolebrutinib 5/60 mg | Tolebrutinib 15/60 mg | Tolebrutinib 30/60 mg | Tolebrutinib 60/60 mg
Number analyzed (Participants) | 31 | 31 | 32 | 31
relapses per participant year | 0.26 [0.15 to 0.46] | 0.24 [0.14 to 0.42] | 0.28 [0.18 to 0.43] | 0.23 [0.13 to 0.38]

6. Secondary Outcome: Change From Baseline in Expanded Disability Status Scale (EDSS) Score at Week 240
Description: The EDSS is a disability scale that assesses the following 7 functional domains: visual, brainstem, pyramidal (motor), cerebellar (coordination), sensory, cerebral, and bowel/bladder. The total EDSS ranges from 0 (normal) to 10 (death due to MS) (0.5 increments from 1-10; next increase after 0 is 1). Higher scores indicated increased disability. Baseline assessed for long-term tolebrutinib treatment by change from baseline was defined as the last non-missing value prior to the first administration of randomized study drug in DRI15928 study.
Time Frame: Baseline (Day 1 of DRI15928) and Week 240
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tolebrutinib 5/60 mg | Tolebrutinib 15/60 mg | Tolebrutinib 30/60 mg | Tolebrutinib 60/60 mg
Number analyzed (Participants) | 21 | 23 | 21 | 26
score on a scale | -0.10 (0.96) | 0.24 (0.95) | 0.38 (0.69) | 0.29 (0.70)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study drug (Day 1) up to maximum exposure, 39 weeks in Part A and 222 weeks in Part B. All-cause mortality (deaths) was collected from signing informed consent form (Week -6) up to end of follow-up, approximately 62 months
Description: Analysis was performed on the safety population.
Arm/Group | Part A: Tolebrutinib 5 mg | Part A: Tolebrutinib 15 mg | Part A: Tolebrutinib 30 mg | Part A: Tolebrutinib 60 mg | Part B: Tolebrutinib 5/60 mg | Part B: Tolebrutinib 15/60 mg | Part B: Tolebrutinib 30/60 mg | Part B: Tolebrutinib 60/60 mg
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31 | 0/32 | 0/31 | 0/30 | 0/31 | 0/32 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 2/31 | 1/32 | 2/31 | 5/30 | 3/31 | 3/32 | 3/31
Other Adverse Events (participants affected / at risk) | 12/31 | 6/31 | 15/32 | 16/31 | 24/30 | 24/31 | 24/32 | 25/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Tolebrutinib 5 mg (N=31) | Part A: Tolebrutinib 15 mg (N=31) | Part A: Tolebrutinib 30 mg (N=32) | Part A: Tolebrutinib 60 mg (N=31) | Part B: Tolebrutinib 5/60 mg (N=30) | Part B: Tolebrutinib 15/60 mg (N=31) | Part B: Tolebrutinib 30/60 mg (N=32) | Part B: Tolebrutinib 60/60 mg (N=31)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Burn Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Infected Bite (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative Wound Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple Sclerosis Relapse (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Uterine Polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint Dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Tolebrutinib 5 mg (N=31) | Part A: Tolebrutinib 15 mg (N=31) | Part A: Tolebrutinib 30 mg (N=32) | Part A: Tolebrutinib 60 mg (N=31) | Part B: Tolebrutinib 5/60 mg (N=30) | Part B: Tolebrutinib 15/60 mg (N=31) | Part B: Tolebrutinib 30/60 mg (N=32) | Part B: Tolebrutinib 60/60 mg (N=31)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 10 (10) | 10 (12) | 7 (9) | 14 (20)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Cystitis Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (7) | 5 (14)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 5 (7) | 6 (11) | 4 (6) | 6 (12)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 4 (4) | 2 (3) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 1 (2) | 4 (4) | 4 (7) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 5 (6) | 3 (5)
Urinary Tract Infection Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 3 (3) | 2 (2) | 3 (3) | 4 (4)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Seasonal Allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Carpal Tunnel Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 4 (4) | 3 (4) | 2 (4) | 1 (2) | 2 (2) | 3 (3)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (4) | 0 (0)
Tension Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 5 (5)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 6 (7) | 5 (7) | 1 (1) | 3 (3)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Renal Colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 0 (0)
Foot Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Influenza Like Illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT03996291/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT03996291/SAP_001.pdf